CLINICAL TRIAL: NCT00630019
Title: Ocular Tissue Levels of 1.5% Levofloxacin Ophthalmic Solution Compared to an Active Comparator
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: Vistakon Pharmaceuticals (Industry)
Responsible Party: Brian Schwam, MD, VISTAKON Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VPH0107
Record Dates: First submitted 2008-02-22; First posted 2008-03-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Cataract
Keywords: Aqueous humor penetration by anti-infectives
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 1.5% levofloxacin ophthalmic solution
- 2 (Active Comparator)
  Interventions: Drug: 0.5% moxifloxacin hydrochloride ophthalmic solution

INTERVENTIONS:
Drug: 1.5% levofloxacin ophthalmic solution — Topical application
  Arms: 1
Drug: 0.5% moxifloxacin hydrochloride ophthalmic solution — Topical application
  Arms: 2

SUMMARY:
Compare ocular tissue levels following topical ocular instillation of 1.5% levofloxacin ophthalmic solution or an active comparator in subjects undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Capable of instilling eye drop
* Scheduled for cataract surgery with intraocular lens (IOL) implantation
* Be medically cleared for surgery
* Women must be postmenopausal (for at least 1 year), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry, and must agree to continue to use the same method of contraception throughout the study
* Women of childbearing potential must have a negative urine pregnancy test at screening.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Subjects (or his/her legally acceptable representative) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Known allergy or other contraindication to the test article(s) or their components.
* Presence of any abnormality or significant illness in the eye that in the investigator's opinion could affect the subject's health or the study parameters.
* History of or presence of any corneal pathology or disease
* Presence of an active ocular infection (bacterial, viral or fungal), or positive history of ocular herpetic infection.
* History of severe dry eye syndrome.
* History or evidence of previous ocular surgery in the operative eye.
* History of any significant illness that could be expected to interfere with the study parameters.
* Use of disallowed therapies (systemic or topical):

  * Fluoroquinolone anti-infective agents (systemic or topical) within 2 weeks of Visit 1 or anytime after Visit 1 for the duration of the study;
  * Topical ophthalmic preparations (including tear substitutes and rewetting drops), within 1 week of Visit 1 or anytime after Visit 1 for the duration of the study (other than the study medication as restricted above), with the exception of non-steroidal topical ophthalmic drops
* Use of contact lenses in the 2 weeks prior to the study and for the duration of the study.
* Received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment.
* Pregnant or breast-feeding.
* Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Concentration of levofloxacin and active control in the aqueous humor | Time of surgery

SECONDARY OUTCOMES:
Adverse Events | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bucci Laser Vision & Ambulatory Surgery Center, Wilkes-Barre, Pennsylvania, United States